CLINICAL TRIAL: NCT00741897
Title: A Monitored Release Study On The Efficacy And Safety of Fexofenadine (Telfast®) 30mg Pediatric Tablets On Filipino Children Aged 6 To 11 for The Relief of Perennial And Intermittent Allergic Rhinitis.
Brief Title: Fexofenadine Study On Filipino Children for The Relief of Perennial And Intermittent Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M016455C_4001
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — fexofenadine

ARMS (1):
- 1 (Experimental): Fexofenadine
  Interventions: Drug: Fexofenadine

INTERVENTIONS:
Drug: Fexofenadine — Fexofenadine: One 30 mg Tablet once daily for two weeks

SUMMARY:
To determine the safety and efficacy of Fexofenadine (Telfast®) 30mg pediatric tablets on Filipino children aged 6 to 11 for the relief of symptoms associated with perennial and intermittent allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Children who manifest allergic rhinitis symptoms such as sneezing, rhinorrhea, itchy nose/palate/throat and/or itchy/watery/red eyes.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Actual)
Dates: Start 2002-03; Primary Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Patient's assessment of symptoms and drug activity (Total symptom scores) | At baseline, D 7 and D 14
Physician's assessment of symptoms and drug activity (Total symptom scores) | At D 14

SECONDARY OUTCOMES:
AE and SAE collection | From the signature of the informed consent up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Pagunsan, Study Director — Sanofi
Locations (1):
- Sanofi-aventis administrative office, Makati City, Philippines